CLINICAL TRIAL: NCT06643507
Title: Clinical Evaluation of the Modified VISTA Technique (M-VISTA )Using Albumin-platelet Rich Fibrin (Alb-PRF) Versus Connective Tissue Graft (CTG)in the Treatment of Multiple Miler Class III RT2 Recessions A Randomized Clinical Trial
Brief Title: Evaluation of the Modified VISTA Technique Using ALB-PRF vs CTG in the Treatment of Multiple Miller Class III Recessions
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamani Mahmoud Abdullah Fakhri, clinical evaluation of the modified VISTA technique (M-VISTA)using Albumin -platelet rich fibrin (Alb-PRF)versus connective tissue graft (CTG)in the treatment of multiple miller class III/RT2recessions : a randomized clinical trial, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER 3 -3 -1
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Gingival Recession
Keywords: gingival recession, plastic surgery, soft tissue management
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with gingival recession control group (Active Comparator): patients with gingival recessions of miller class III /RT2 the control group will be treated with modified vista technique using connective tissue graft
  Interventions: Other: Connective tissue graft
- patients with gingival recession interventional group (Experimental): patients with gingival recessions of miller class III /RT2 the interventional group will be treated with modified vista technique using albumin PRF
  Interventions: Biological: ALB-PRF

INTERVENTIONS:
Other: Connective tissue graft — regenerative properties
  Arms: patients with gingival recession control group
Biological: ALB-PRF — regenerative properties
  Arms: patients with gingival recession interventional group

SUMMARY:
treatment of miller class III RT2 gingival recession using modified vista technique using connective tissue graft vs albumin PRF

DETAILED DESCRIPTION:
treatment of gingival recession is an important element in the treatment of periodontitis this study covers clinical evaluation of using the modified VISTA technique with using Albumin-PRF VS connective tissue graft in the treatment of miller class III / RT2 for root coverage outcomes

ELIGIBILITY:
Inclusion Criteria:

* 18 years old good oral hygiene

Exclusion Criteria:

* smokers patients with poor oral hygiene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
mean root coverage | 6 months
  primary outcome measures of mean root coverage in millimeters by UNC15 periodontal probe

SECONDARY OUTCOMES:
the percentage of mean root coverage | 6 months
  secondary outcome measures in percentage by UNC15 probe
the percentage of complete root coverage | 6 months
  measures in percentage by using UNC periodontal probe
recession depth | 6 months
  measures in millimeters by using UNC15 periodontal probe
recession width | 6 months
  measures in millimeters by using UNC 15periodontal probe
keratinized tissue width | 6 months
  measures in millimeters by using UNC15 periodontal probe
clinical attachment level | 6 months
  measures by millimeters by using UNC 15 periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Enji EA Ahmed, BDS.MDS.PHD, Study Director — Cairo University; Sarah SE Elbanna, BDS.MDS.PHD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt